CLINICAL TRIAL: NCT06094283
Title: Double-blind, Placebo Controlled, First in Human Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Oral Doses of YCT-529
Brief Title: First in Human Study Evaluating Single Ascending Oral Doses of YCT-529 in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: YourChoice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: YCT-529-01; 1007466 (Other: IRAS)
Record Dates: First submitted 2023-05-03; First posted 2023-10-23 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Male Contraception
Keywords: male; non-hormonal; male contraception; healthy males; sperm count reduction; sperm motility; impaired spermatogenesis; impaired motility; orally administered; vasectomy; vasectomized men

STUDY DESIGN:
Intervention Model Description: In each cohort, the first 2 sentinel subjects will be randomized in a 1:1 ratio to receive either YCT-529 or placebo. The remaining 6 subjects in each cohort will be enrolled in the dosing cohort such that 5 subjects will be randomized to receive YCT-529 and 1 subject will be randomized to receive placebo; therefore, a total of 6 subjects will be randomized to receive YCT-529 and 2 subjects will be randomized to receive placebo at each dose level.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind, placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- YCT-529 (Active Comparator): Oral single ascending dose(s)
  Interventions: Drug: YCT-529
- Placebo (Placebo Comparator): Placebo for YCT-529 Capsule
  Interventions: Drug: YCT-529 Placebo

INTERVENTIONS:
Drug: YCT-529 — Single oral dose (planned doses of 10, 30, 90 and 200 mg; dose levels will not exceed 250 mg
  Arms: YCT-529
Drug: YCT-529 Placebo — YCT-529 Placebo
  Arms: Placebo

SUMMARY:
A single ascending oral dose(s) study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of YCT-529 in healthy male subjects.

DETAILED DESCRIPTION:
This is a Phase 1a, double-blind, placebo controlled, first in human study to evaluate the safety, tolerability, PK, and PD of YCT-529 in 2 cohorts of 8 subjects. Cohorts 1 and 2 will be dosed in the fasted state in Periods 1 and 2. Each cohort will receive two doses of study drug separated by a washout period. One cohort will then return for a third dose of study drug under fed conditions in Period 3 to study the effect of food on YCT-529.

ELIGIBILITY:
Inclusion Criteria:

1. Male subject in good health as confirmed by physical examination, medical history, and clinical laboratory tests of blood and urine at the time of Screening.
2. Subject must provide written informed consent.
3. Subject must be willing and able to communicate and participate in the whole study.
4. Subject is 25 to 60 years of age (inclusive).
5. Subject has been vasectomized for at least 6 months prior to enrolment
6. Subject has body mass index (BMI) 18.0 to 32.0 kg/m2.
7. Subject has no history of hormonal therapy uses in the 90 days prior to the first screening visit.
8. Subject agrees to use a condom during the study until the final return visit to ensure the safety of the study participants and their sexual partner(s)
9. Subjects will refrain from donating blood or plasma during the study.
10. Subjects will not use cannabis or any recreational drugs for at least 120 days before completing Screening and during the study.
11. In the opinion of the investigator, subject is able to adhere to the study requirements, restrictions, schedule of assessments, and requirements related to sperm sample collection and maintenance of the sexual activity diary.

Exclusion Criteria:

1. Men participating in another clinical study involving an investigational drug within the last 90 days prior to the first dosing or less than 5 elimination half-lives prior to first dosing, whichever is longer.
2. Clinically significant abnormal physical and/or laboratory findings at Screening
3. Abnormal serum chemistry values at screening or admission, that indicate liver or kidney dysfunction or that may be considered clinically significant, such as bilirubin of >20 micro mol/L and ALT, AST, GGT and ALP above the upper limit of normal.
4. Evidence of renal impairment at screening, as indicated by an estimated eGFR of <80 mL/min/1.73 m2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI; 2009) equation.
5. Use of androgens within 90 days before first screening visit.
6. Ongoing use of body building nutritional supplements.
7. Systolic blood pressure (BP) >140 mmHg (<45 years) or >160 mmHg (≥45 years) and diastolic BP >90 mmHg at screening or predose.
8. Clinically significant abnormal electrocardiogram (ECG) or a duration of corrected QT interval in ECG (QTc) interval of >450 msec at screening or predose.
9. Known history of androgen deficiency due to hypothalamic-pituitary or testicular disease or multiple endocrine deficiencies.
10. Known history of significant cardiovascular, renal, hepatic (cholecystectomy is not permitted), or prostatic disease or significant psychiatric illness. Gilbert's syndrome is allowed (subject will be excluded if total bilirubin is ≥1.5 x ULN if known Gilbert's syndrome). If subject has elevations only in total bilirubin that are >ULN and <1.5xULN, fractionate bilirubin to identify possible undiagnosed Gilbert's syndrome (i.e., direct bilirubin <35% of the total bilirubin).
11. Current or clinically relevant history of any psychiatric disorder or clinical assessment of significant suicidal risk or risk of self-injury as per the Investigator's judgement. This will be re-assessed at admission to Period 2 and Period 3 if applicable.
12. Serious adverse reaction or serious hypersensitivity to any drug or formulation excipients.
13. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active.
14. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) 1 and 2 antibody results at screening visit.
15. Known or suspected alcoholism or drug abuse within the last 2 years that may affect metabolism/transformation of steroid hormones or study treatment compliance.
16. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator or delegate at screening.
17. Regular alcohol consumption in males >14 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type).
18. Current smokers and those who have smoked within the last 6 months. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission.
19. Confirmed positive drugs of abuse test result.
20. Subjects who are taking, or have taken, any prescribed or over-the-counter drug or vitamins/herbal remedies/supplements (other than up to 4 g of paracetamol per day in the 14 days before IMP administration). COVID-19 vaccines are accepted concomitant medications. Exceptions may apply, as determined by the investigator, if each of the following criteria are met: medication with a short half-life if the washout is such that no PD activity is expected by the time of dosing with IMP; and if the use of medication does not jeopardize the safety of the trial subject; and if the use of medication is not considered to interfere with the objectives of the study.
21. Male subjects with pregnant or lactating partners.
22. Subjects who are taking, or have taken, any prescribed or over-the-counter drug or vitamins/herbal remedies/supplements (other than up to 4 g of paracetamol per day in the 14 days before IMP administration). COVID-19 vaccines are accepted concomitant medications. Exceptions may apply, as determined by the investigator, if each of the following criteria are met: medication with a short half-life if the washout is such that no PD activity is expected by the time of dosing with IMP; and if the use of medication does not jeopardize the safety of the trial subject; and if the use of medication is not considered to interfere with the objectives of the study.
23. Any site staff member with delegated study responsibilities or a family member of a site staff member with delegated study responsibilities.
24. Any other medical condition that, in the opinion of the investigator, could alter the subject's well-being, the study conduct, or the interpretability of the results.

    -

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Sex assigned at birth is required to be "male"
Enrollment: 16 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
The incidence and nature of any adverse events, dose-limiting adverse events and serious adverse adverse events. | Baseline to 43 days for subjects participating in Cohorts 1 and 2 participating in the 2 periods; Baseline to 10 weeks for Cohorts 1 and 2 that also complete the fed portion of the study; and Baseline to 16 weeks if waiting for other cohorts to finish
  Assessment of the number and type of adverse events, dose-limiting adverse events and serious adverse events following dosing.
Vital signs assessment (heart rate) | Baseline to Day 15
  Changes from pre-dose values (beats per minute)
Vital signs assessment (blood pressure) | Baseline to Day 15
  Changes from pre-dose values (mm hg)
Vital signs assessment (oral temperature) | Baseline to Day 15
  Changes from pre-dose values (temperature in celsius degrees)
12-lead ECG assessment (heart rate) | Baseline to Day 15
  Changes from pre-dose values (beats per minute)
12-lead ECG assessment (QT interval) | Baseline to Day 15
  Changes from pre-dose values for QT internal length (msec)
12-lead ECG assessment (QTcF Interval) | Baseline to Day 15
  Changes from pre-dose values for QTcF interval length (msec)
12-lead ECG assessment (PR Interval) | Baseline to Day 15
  Changes from pre-dose values for PR interval length (msec)
12-lead ECG assessment (QRS Duration) | Baseline to Day 15
  Changes from pre-dose values for QRS duration (msec)
Clinical laboratory assessments (hematology blood sample tests) | Baseline to Day 15
  Changes from pre-dose values (Tests: Hemoglobin, Hematocrit, packed cell volume, Red blood cell, erythrocyte count, mean corpuscular volume, mean corpuscular hemoglobin, Mean corpuscular hemoglobin concentration, Platelet count, White blood cell, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils
Clinical laboratory assessments (coagulation blood sample tests) | Baseline to Day 15
  Changes from pre-dose values (Tests: Prothrombin time, Activated partial thromboplastin time (APTT), Fibrinogen)
Clinical laboratory assessments (clinical chemistry blood sample tests) | Baseline to Day 15
  Changes from pre-dose values (Tests: Sodium, Potassium, Chloride, Bicarbonate, Urea, Creatinine, Bilirubin (total), Bilirubin (direct; only if total is elevated), Alkaline phosphatase, Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Lactate dehydrogenase (LDH), Creatine kinase (CK), Gamma glutamyl transferase (GGT), Protein (Total), Albumin, Calcium, Glucose (fasting), Glucose,Triglycerides (fasting) Cholesterol (total; fasting)
Clinical laboratory assessments (urine sample tests) | Baseline to Day 15
  Changes from pre-dose values (Bilirubin, Urobilinogen, Ketones, Glucose, Protein, Blood, Nitrites, pH, Specific gravity, Leukocytes)

SECONDARY OUTCOMES:
Plasma PK Parameter of YCT-529 (Area under the curve to Infinity [AUCinf]) | Pre-dose to 336 hours after dosing
  Plasma PK Parameter as measured by area under the curve from time 0 extrapolated to infinity [AUCinf],
Plasma PK Parameter of YCT-529 (Area under the curve to the last measured concentration [AUC0-t]) | Pre-dose to 336 hours after dosing
  Plasma PK Parameter as measured by area under the curve from time 0 to the last measured concentration [AUC0-t]
Plasma PK Parameter of YCT-529 (Area under the curve to 24 hours [AUC0--24]) | Pre-dose to 336 hours after dosing
  Plasma PK Parameter as measured by area under the curve from time 0 to 24 hours [AUC0--24]
Plasma PK Parameter of YCT-529 (Time to maximum concentration [Tmax]) | Pre-dose to 336 hours after dosing
  Plasma PK Parameter as measured by time to maximum concentration [Tmax]
Plasma PK Parameter of YCT-529 (Terminal elimination half life [T1/2]) | Pre-dose to 336 hours after dosing
  Plasma PK Parameter as measured by terminal elimination half life [T1/2]
Plasma PK Parameter of YCT-529 (Lag time [Tlag]) | Pre-dose to 336 hours after dosing
  Plasma PK Parameter as measured by lag time [Tlag]
Plasma PK Parameter of YCT-529 (Volume of distribution [Vz/F]) | Pre-dose to 336 hours after dosing
  Plasma PK Parameter as measured by apparent volume of distribution [Vz/F]
Plasma PK Parameter of YCT-529 (oral clearance [CL/F]) | Pre-dose to 336 hours after dosing
  Plasma PK Parameter as measured by oral clearance [CL/F] of YCT-529, including the effect of food on the PK
Plasma PK Parameter of YCT-529 (maximum concentration [Cmax]) | Pre-dose to 336 hours after dosing
  Plasma PK Parameter as measured by maximum concentration [Cmax]) of YCT-529, including the effect of food on the PK
Pharmacodynamic parameter of YCT-529, including follicle-stimulating hormone | Pre-dose to 336 hours after dosing
  Changes from pre-dose values of follicle-stimulating hormone
Pharmacodynamic parameter of YCT-529, including luteinizing hormone | Pre-dose to 336 hours after dosing
  Changes from pre-dose values of luteinizing hormone
Pharmacodynamic parameter of YCT-529, including testosterone | Pre-dose to 336 hours after dosing
  Changes from pre-dose values of testosterone
Pharmacodynamic parameter of YCT-529, including sex hormone binding globulin | Pre-dose to 336 hours after dosing
  Changes from pre-dose values of including sex hormone binding globulin

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, MBChB, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Nottingham, East Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mannowetz N, McCallum SW, Sidhu S, Mena KH, Ruby EP, Castro-Santamaria R, Dodds E, Henderson D, Whitaker G, Wright H, Beaudoin S, Bakshi A. Safety and pharmacokinetics of the non-hormonal male contraceptive YCT-529. Commun Med (Lond). 2025 Jul 22;5(1):279. doi: 10.1038/s43856-025-01004-4. PMID 40696162